CLINICAL TRIAL: NCT02427308
Title: Treatment of Leishmaniasis With Impavido® (Miltefosine): Pregnancy Registry
Status: Withdrawn | Type: Observational
Why Stopped: Study completed and no patients registered
Sponsor: Knight Therapeutics (USA) Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: IMP 2127-1
Record Dates: First submitted 2015-04-22; First posted 2015-04-28 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Leishmaniasis or Other Uses of Miltefosine
Keywords: leishmaniasis; miltefosine; pregnancy
MeSH Terms: conditions — Leishmaniasis | interventions — miltefosine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- miltefosine patients that become pregnant
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine — target dose = 2.5 mg/kg/day for 28 days

SUMMARY:
The purpose of this observational study is to fulfill FDA Post Marketing Requirement (PMR) 2127-1 for miltefosine (NDA204684): implement a pregnancy registry for the time period Mar 2015-Mar 2024.

This study is a prospective observational study in which female patients undergoing Impavido who become pregnant during treatment or within 5 months after completing treatment can volunteer to provide information about their pregnancy and the outcome of the pregnancy.

DETAILED DESCRIPTION:
Objective: The purpose of this observational study is to fulfill FDA Post Marketing Requirement (PMR) 2127-1 for miltefosine (NDA204684): implement a pregnancy registry for the time period Mar 2015-Mar 2024.

Study Design: This study is a prospective observational study in which female patients undergoing Impavido who become pregnant during treatment or within 5 months after completing treatment can volunteer to provide information about their pregnancy and the outcome of the pregnancy. Information will be collected from patient's provider of Impavido treatment, obstetrical treatment, and if applicable, the child's pediatrician.

Population: Leishmaniasis patients or patients who take Impavido off-label who become pregnant while taking Impavido or within 5 months after taking Impavido.

Drug Product:

Drug name: Impavido (50 mg capsules). Dosing regimen: as per the Impavido Product Label (PL)

Study Procedures: Pregnant women will become aware of the Impavido Pregnancy Registry via the product label (PL) or the Impavido website or her physician. By calling 1-866-588-5405, the patient will be connected to the Impavido Pregnancy Registry Coordinating Center. A trained staff member will acquaint the patient with the goals and procedures of the study. If the patient tentatively agrees to participate in the study over the telephone, the patient will be mailed information forms, the Consent Form and Assent Form as appropriate, and the Consent for the patient's physician and obstetrician and the child's pediatrician to release medical information. Receipt of the four signed Consent Forms and Assent Form as appropriate by the Coordinating Center will signify patient and/or legal guardian consent/assent. The Coordinating Center will contact the patient and/or the patient's physicians each trimester until delivery to collect data on maternal adverse events (AEs), pregnancy outcome, and fetal outcome.

Sample Size And Study Duration: Estimated 0-1 patients per year for 10 years.

Outcome Parameters:

Maternal AEs. Pregnancy outcome. Fetal outcome.

Analysis Plan: Baseline data, compliance to prescribed treatment, and outcomes will be reported for individual patients and for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Has the subject received Impavido?
2. Is the subject a female?
3. Did the subject become pregnant during Impavido treatment or within 5 months after completing treatment?
4. Did the subject or legal guardian give consent/assent for the study and to collect data from her physicians?

Exclusion Criteria:

[none]

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: persons who become pregnant will taking miltefosine or for 5 months after taking miltefosine
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
number of patients with adverse effects during pregnancy | 9 months
number of patients with adverse pregnancy outcome | 9 months
number of patients with adverse fetal outcome | at birth

CONTACTS AND LOCATIONS:
Overall Officials: Janet Ransom, PhD, Principal Investigator — Fast Track Drugs and Biologics LLC
Locations (1):
- Fast Track, North Potomac, Maryland, United States